CLINICAL TRIAL: NCT05389423
Title: Phase I Trial of Pomalidomide and Dose-Adjusted EPOCH +/- Rituximab for HIV-Associated Lymphomas
Brief Title: Pomalidomide and Dose-Adjusted EPOCH +/- Rituximab for HIV-Associated Lymphomas
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 10000274; 000274-C
Record Dates: First submitted 2022-05-21; First posted 2022-05-25 (Actual); Last update posted 2025-06-24 (Actual); Status verified 2025-06-16

CONDITIONS: Diffuse Large Cell Lymphoma; Non-Hodgkin Lymphoma; Burkitt Lymphoma; Plasmablastic Lymphoma; B-Cell Neoplasm
Keywords: Non-Hodgkin Lymphoma; Epstein Barr Virus; Plasmablastic Lymphoma; Chemotherapy; Immune Modulatory
MeSH Terms: conditions — Lymphoma, Large B-Cell, Diffuse; Lymphoma, Non-Hodgkin; Burkitt Lymphoma; Plasmablastic Lymphoma; Lymphoma, B-Cell; Epstein-Barr Virus Infections | interventions — Vincristine; Prednisone; Doxorubicin; Etoposide; pomalidomide; Cyclophosphamide; Rituximab

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- 1/Dose Escalation (Experimental): Pomalidomide (escalating doses) + Prednisone, Etoposide, Doxorubicin, Vincristin
  Interventions: Drug: Vincristine; Drug: Prednisone; Drug: Doxorubicin; Drug: Etoposide; Drug: Pomalidomide; Drug: Cyclophosphamide; Drug: Rituximab
- 2/Dose Expansion (Experimental): Pomalidomide (at the MTD) + Prednisone, Etoposide, Doxorubicin, Vincristine and
  Interventions: Drug: Vincristine; Drug: Prednisone; Drug: Doxorubicin; Drug: Etoposide; Drug: Pomalidomide; Drug: Cyclophosphamide; Drug: Rituximab

INTERVENTIONS:
Drug: Vincristine — 0.4 mg/m2/day administered by CIVI on days 1 to 4
Drug: Prednisone — 60 mg/m2/day administered orally on days 1 to 5
Drug: Doxorubicin — 10 mg/m2/day administered by CIVI on days 1 to 4
Drug: Etoposide — 50 mg/m2/day administered by CIVI on days 1 to 4
Drug: Pomalidomide — An initial dose of 3mg administered orally for 10 days in all cycles. In cycle 1, it will start 5 days before DA-EPOCH; in cycles 2-6, it will start on day 1. Administered at an MTD dose for the expansion phase.
Drug: Cyclophosphamide — 750 mg/m2 administered IV on day 5
Drug: Rituximab — 375 mg/m2 administered IV on day 1 (only for CD20+ tumors)

SUMMARY:
Background:

Non-Hodgkin lymphoma (NHL) is the most common cancer among people living with HIV in the United States. People with HIV are up to 17 times more likely to get NHL than people who do not have HIV. The disease may also be different in these two groups. More study is needed for treating

people with both HIV and NHL.

Objective:

To test a study drug (pomalidomide) in combination with chemotherapy with or without another drug (rituximab) in people with HIV-associated NHL.

Eligibility:

Adults aged 18 years or older diagnosed with HIV-associated B-cell NHL with high-risk features.

Design:

Individuals will undergo screening. They will have a physical exam. They will have blood and urine tests and tests of heart function. They may have imaging scans. Researchers will review tissue samples of individual s tumors. In some cases, a new biopsy may be needed.

Individuals will receive up to 6 cycles of treatment.

The first cycle is 26 days: Individuals will take pomalidomide by mouth for 10 days. After 5 days they will start receiving chemotherapy drugs through a tube attached to a needle placed in a vein (IV). Some participants will receive rituximab on day 5. All individuals will receive a second set of IV drugs that will last for 4 days (96 hours). They will receive another IV drug after the previous treatment is complete.

The remaining cycles are each 21 days. Individuals will take pomalidomide by mouth for the first 10 days. Other chemotherapy treatments will also be repeated starting on day 1 of each cycle.

Screening tests will be repeated at study visits.

Follow-up visits will continue for 4 years....

DETAILED DESCRIPTION:
Background:

* Non-Hodgkin lymphoma (NHL) is the most common cancer among people living with human immunodeficiency virus (HIV) (PLWH) in the United States. Even in the modern era of antiretroviral therapy (ART), PLWH have an 11- to 17-fold higher risk of NHL than the general population due in part to CD4+ T-cell lymphopenia but also immune dysregulation and exhaustion from chronic viral antigen stimulation.
* The most common NHL subtypes are diffuse large cell lymphoma (DLBCL) and Burkitt lymphoma (BL), that are much more frequently associated with the oncogenic virus Epstein Barr virus (EBV) in PLWH, which portends a poorer prognosis, than in the general population.
* Plasmablastic lymphoma (PBL) is a rare CD20 negative B cell lymphoma associated with EBV almost exclusively seen in PLWH.
* Although these subtypes of lymphoma occur in the general population, their presentation and pathogenesis may be different - meaning there may be different therapeutic targets and strategies to consider in HIV-associated lymphomas necessitating clinical trials targeted to this underserved population of patients.
* Lenalidomide, a 2nd generation immunomodulatory drug, has shown safety and improved survival in combination with chemotherapy in advanced stage DLBCL in one of two randomized trials.
* Pomalidomide, a 3rd generation immunomodulatory agent, has activity in primary central nervous system (CNS) lymphoma demonstrating its activity in both NHL and CNS involvement, which is more common in PLWH and NHL. In a number of parameters, it is more potent than lenalidomide.
* Pomalidomide has shown to increase natural killer (NK) and T-cell activation and reverse T-cell senescence in addition to increasing CD4+ T-cell count in PLWH and cancer. It can also enhance expression of surface immune markers in vitro in cell lines from EBV-induced tumors.
* Dose-adjusted etoposide, prednisone, vincristine, cyclophosphamide, and doxorubicin (DA-EPOCH) along with rituximab (DA-EPOCH-R) is an anthracycline-based regimen that has been shown to be safe and effective in PLWH and in the most common subtypes of NHL seen in PLWH, DLBCL and BL.

Objective:

-Determine the safety and maximum tolerated dose (MTD) of the combination of pomalidomide and dose-adjusted EPOCH +/ rituximab (DA-EPOCH-RP) in participants with enrolled subtypes of HIV-associated lymphomas

Eligibility:

* Adult participants >= 18 years with pathology-confirmed HIV-associated B-cell non-Hodgkin lymphoma with high-risk features, excluding primary CNS lymphoma
* Positive HIV1/2 serology

Design:

* This is a phase 1 study of DA-EPOCH-RP in participants with HIV-associated B-cell non-Hodgkin lymphoma. Only participants with CD20+ HIV-associated B-cell non-Hodgkin lymphoma will receive Rituximab.
* This is a dose escalation study to evaluate pomalidomide in combination with modified DA-EPOCH-R to determine safety and tolerability. Dosing will begin at dose level 1, 3 mg of pomalidomide and proceed to dose escalation or de-escalation to doses 4 mg or 2 mg depending on dose-limiting toxicities.
* Participants will be prescribed ART.
* In this phase I study, up to 12 evaluable participants will be accrued in the escalation phase (3-6 participants per level) and up to 6 evaluable participants will be accrued in the expansion phase to be treated at MTD.

ELIGIBILITY:
* INCLUSION CRITERIA:
* Histologically or cytologically confirmed B-cell NHL confirmed by the Laboratory of Pathology (LP), NCI, with one or more of the following features:

  * Leptomeningeal/CSF involvement
  * High-risk for CNS relapse per CNS-IPI (score 4-6)
  * Plasmablastic histology
  * Gamma herpesvirus positive tumor
  * Presence of KS
* Measurable or evaluable lymphoma.
* Positive HIV1/2 serology.
* Individuals may not have received prior curative-intent chemotherapy for lymphoma. Individuals who have received prior treatment as a bridge to curative-intent therapy will be considered per Protocol Chair discretion if >= 2 weeks since administration. Steroids given for any reason or rituximab given for multicentric Castleman disease may be given any time prior to treatment start.
* Age >=18 years
* Eastern Cooperative Oncology Group performance status (ECOG-PS) <=4
* Individuals of childbearing potential (IOCBP) must have a negative serum or urine pregnancy test with a sensitivity of at least 25 mIU/mL within 2 weeks prior to and again within 1 day before starting the study drugs and must either commit to continued abstinence from penetrative vaginal intercourse or begin TWO acceptable methods of birth control, one highly effective method and one additional effective method AT THE SAME TIME, at least 28 days before the participant starts taking pomalidomide and for 12 months after the last dose of combined chemotherapy.
* Individuals able to father a child must agree to use an effective method of contraception (barrier, surgical sterilization, abstinence) for the duration of the study treatment and up to six (6) months after the last dose of the study drug(s). We also will recommend individuals able to father a child with IOCBP partners to ask the partners to be on an effective birth control (hormonal, intrauterine device (IUD), surgical sterilization). Individuals able to father a child must not freeze or donate sperm within the same period.
* All individuals must agree to be registered into the mandatory POMALYST REMS(R)TM program and be willing and able to comply with the requirements of the POMALYST REMS(R)TM program.
* Able to take aspirin 81mg orally daily or another substitute thromboprophylaxis.
* Adequate organ and marrow function as defined below unless abnormalities are attributed to lymphoma or HIV as determined by investigator:

  * absolute neutrophil count >=1,000/mcL
  * platelets >=75,000/mcL
  * total bilirubin <=1.5 X institutional upper limit of normal (individuals with history of Gilbert disease are eligible if total bilirubin <= 5 mg/dL with <80% unconjugated bilirubin)
  * aspartate aminotransferase (AST) / alanine transaminase (ALT) <=3 X institutional upper limit of normal
  * creatinine clearance >=60 mL/min/1.73 m^2 for individuals with creatinine levels above institutional normal.
* Hepatitis B virus (HBV) infection must be on suppressive antiviral therapy.
* Willingness to take and adhere to ART (individuals are not required to be on any specific regimen of ART).
* Individuals must understand and sign a written informed consent document.

EXCLUSION CRITERIA:

* Individuals may not receive investigational agents on other clinical trials.
* Requirement of any of the agents listed as prohibited thearapies.
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to pomalidomide or other agents used in study.
* Parenchymal brain involvement with lymphoma.
* Ejection fraction less than 40% by echocardiography (ECHO)
* CTCAEv5.0 Grade 3-4 neuropathy
* History of malignant tumors other than KS or KSHV-associated multicentric Castleman Disease, (MCD), unless:

  * In complete remission for >= 1 year from the time response was first documented; or,
  * Completely resected basal cell carcinoma; or,
  * In situ squamous cell carcinoma of the cervix or anus; or,
  * Prior or concurrent malignancy has a natural history or treatment which does not have the potential to interfere with the safety or efficacy assessment of the investigational regimen per Protocol Chair discretion.
* Known drug-related, inherited, or acquired procoagulant disorder including prothrombin gene mutation 20210, antithrombin III deficiency, protein C deficiency, protein S deficiency and antiphospholipid syndrome but not including heterozygosity for the Factor V Leiden mutation or the presence of a lupus anticoagulant in the absence of other criteria for the antiphospholipid syndrome.
* Symptomatic congestive heart failure
* Unstable angina pectoris, symptomatic cardiac arrhythmia, or cardiac arrhythmia requiring medical treatment.
* Uncontrolled intercurrent illness or participants considered to be of poor medical health due to a serious, uncontrolled medical disorder, non-malignant systemic disease or active uncontrolled infection (excluding lymphoma or HIV) as documented in prior records or suggested by medical history, physical examination or standard clinical assessments such as imaging and laboratory studies.
* Pregnant or nursing individuals (if lactating, must agree not to nurse while taking pomalidomide).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Estimated)
Dates: Start 2023-06-27 (Actual); Primary Completion 2028-06-01 (Estimated); Study Completion 2032-06-01 (Estimated)

PRIMARY OUTCOMES:
safety and tolerability | 6 cycles of treatment, or until confirmed progression, unacceptable toxicity or trial withdrawal
  The fraction of individuals with toxicity noted at each dose level will be reported by grade and type of toxicity identified. Maximum tolerated dose will also be reported.

SECONDARY OUTCOMES:
progression-free survival | every 3 weeks for the first 6 cycles, every 3 months for the rest of the first year, then every 6 months for 4 years (5 years total).
  duration of time from the start of the treatment until time of disease relapse from PR, disease progression, or death, whichever occurs first
preliminary estimates of response | every 3 weeks for the first 6 cycles, every 3 months for the rest of the first year, then every 6 months for 4 years (5 years total).
  Percentage of individuals with the best overall response of CR or PR to therapy

CONTACTS AND LOCATIONS:
Overall Officials: Ramya M Ramaswami, M.D., Principal Investigator — National Cancer Institute (NCI)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: Yes
All IPD recorded in the medical record will be shared with intramural investigators upon request.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Clinical data available during the study and indefinitely.
Access Criteria: Clinical data will be made available via subscription to BTRIS and with the permission of the study PI.

REFERENCES:
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?A_000274-C.html